CLINICAL TRIAL: NCT01932593
Title: Repeat Infusion of Autologous Bone Marrow Cells in Multiple Sclerosis (SIAMMS-II)
Brief Title: Repeat Infusion of Autologous Bone Marrow Cells in Multiple Sclerosis
Acronym: SIAMMS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Bristol NHS Trust (Other)
Collaborators: Sir Halley Stewart Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SIAMMS-II
Record Dates: First submitted 2013-08-13; First posted 2013-08-30 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; bone marrow; stem cell therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: autologous bone marrow cells
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infusion of autologous bone marrow (Experimental): Bone marrow harvest under general anaesthetic and intravenous infusion of filtered but otherwise unselected autologous bone marrow
  Interventions: Procedure: Infusion of autologous bone marrow
- Placebo (Placebo Comparator)
  Interventions: Procedure: Infusion of autologous bone marrow

INTERVENTIONS:
Procedure: Infusion of autologous bone marrow — Bone marrow harvest under general anaesthetic and intravenous infusion of filtered but otherwise unselected autologous bone marrow

SUMMARY:
There is no cure for Multiple Sclerosis (MS) and we are always looking at new ways to stop the disease process and/or promote repair.

We hypothesise that autologous bone marrow cellular therapy in chronic MS offers durable benefit.

The purpose of this study is to test the safety of repeated bone marrow stem cell infusion in patients with MS. We want to find out what effects, good and/or bad, it has on you and your disability.

You have previously participated in a safety study of bone marrow stem cell infusion in patients with MS. The results raised the possibility of some early partial repair; measurements of the speed of neurological impulses in the brain and spinal cord improved. The current study seeks to determine whether those benefits have persisted and whether they can be repeated or enhanced by repeating the procedure.

DETAILED DESCRIPTION:
On the background of our own and others' experimental BM stem cell studies, we recently completed a phase 1 feasibility/safety trial of BM cell therapy in 6 patients with longstanding progressive MS (www.nature.com/clpt/journal/v87/n6/full/clpt201044a.html). Safety was confirmed, and intensive serial neurophysiological tests showed statistically significant improvements at 12 months. While highly preliminary and entirely uncontrolled, these results at least raise the possibility of a beneficial effect within the damaged central nervous system (CNS). A phase 2 clinical trial to formally assess efficacy of intravenous infusion of autologous bone marrow cells in progressive MS will commence in the near future (ACTiMuS trial). This trial comprises a programme of translational and clinical stem cell research, aiming (1) to continue translation with a phase two controlled trial of autologous bone marrow cells (BMCs) in chronic MS; and (2) to explore in parallel the potential mechanisms of action by studying BM cells from treated patients and controls, aiming to establish which BM sub-population(s) contribute(s) to efficacy, and which reparative mechanism(s) are important.

It is not known whether repeated infusion of autologous bone marrow offers additional benefit or how long improvements might be expected to last. The current proposal seeks to explore whether the neurophysiological improvements observed in the phase I study persist several years after the initial single infusion and whether these can be either replicated or augmented by an additional infusion of autologous bone marrow cells.

Hypothesis and aims

We hypothesise that intravenously-delivered autologous bone marrow cellular therapy (BMCT) in chronic MS offers significant benefit. We hypothesize also that the mechanisms are multiple, and include immunomodulation and reparative and/or neuroprotective effects within the CNS; and are offered by one or more BM stem cell sub-populations, jointly contributing to the therapeutic impact. Exploring and understanding these mechanisms, and the biology of the cells responsible, will allow the development of more effective reparative cell therapy in MS.

The current study seeks to examine whether the observed improvements noted in conduction times in central nervous system pathways in the phase I 'Study of Intravenous Autologous Marrow in Multiple Sclerosis (SIAMMS)' persist several years following the initial single infusion and whether these can be either replicated or augmented by an additional infusion of autologous bone marrow cells and analysis of research samples will be performed as per samples included in the concurrent phase 2 clinical trial 'Assessment of bone marrow-derived cellular therapy in progressive multiple sclerosis (ACTiMuS)' (REC 12/SW/0358, ISRCTN27232902, NCT01815632).

ELIGIBILITY:
Inclusion Criteria:

Participation in the phase I safety and feasibility 'Study of Intravenous Autologous Marrow in Multiple Sclerosis' (SIAMMS) (REC reference number number 05/Q1704/137 Clin Pharmacol Ther. 2010 Jun;87(6):679-85)

Exclusion Criteria:

* pregnancy, breastfeeding or lactation
* bone marrow insufficiency
* history of lymphoproliferative disease or previous total lymphoid irradiation immune deficiency
* history of current or recent (<5 years) malignancy
* chronic or frequent drug-resistant bacterial infections or presence of active - infection requiring antimicrobial treatment
* frequent and/or serious viral infection
* systemic or invasive fungal disease within 2 years of entry to study
* significant renal, hepatic, cardiac or respiratory dysfunction
* contraindication to anaesthesia
* bleeding or clotting diathesis
* current or recent (within preceding 12 months) immunomodulatory therapy other than corticosteroid therapy
* treatment with corticosteroids within the preceding 3 months
* radiation exposure in the past year other than chest / dental x-rays
* previous claustrophobia
* the presence of any implanted metal or other contraindication to MRI participation in another experimental study or treatment within previous 24 months

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Adverse events | 1 year post-infusion of autologous bone marrow
  Number of adverse events

SECONDARY OUTCOMES:
Global evoked potential | Baseline then 6 months and 12 months post-infusion of autologous bone marrow
  The 'global evoked potential (GEP)' has been developed as a tool that, by combining multimodal evoked potential recordings to a single score, may be used to monitor the evolution of MS in individual patients, and as a surrogate end point in clinical trials.
MRI brain | Baseline and 6 months post-infusion of autologous bone marrow
  MRI brain scan
Expanded disability status scale (EDSS) | Baseline then 6 months and 12 months post-infusion of autologous bone marrow
  Expanded disability status scale - clinical scale of disability used in MS trials
Multiple sclerosis functional composite (MSFC) | Baseline then 6 months and 12 months post-infusion of autologous bone marrow
  The MSFC is a three-part quantitative assessment of disability and includes a timed walk, the nine-hole peg test and the Paced Auditory Serial Addition Test (PASAT).
Multiple sclerosis impact scale (MSIS-29) | Baseline then 6 months and 12 months post-infusion of autologous bone marrow
  Self-reporting questionnaire re impact of MS

OTHER OUTCOMES:
Tolerability | Ongoing post-infusion of autologous bone marrow with a formal request for feedback at 12 months
  Participants will be encouraged to report their experience of the procedure at any time and to submit a written statement at 12 months post-infusion of autologous bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Neil J Scolding, PhD FRCP, Principal Investigator — North Bristol NHS Trust and University of Bristol
Locations (1):
- North Bristol NHS Trust, Bristol, Avon, United Kingdom

REFERENCES:
- [Derived] Rice CM, Marks DI, Walsh P, Kane NM, Guttridge MG, Redondo J, Sarkar P, Owen D, Wilkins A, Scolding NJ. Repeat infusion of autologous bone marrow cells in multiple sclerosis: protocol for a phase I extension study (SIAMMS-II). BMJ Open. 2015 Sep 11;5(9):e009090. doi: 10.1136/bmjopen-2015-009090. PMID 26363342